CLINICAL TRIAL: NCT05784571
Title: Assessment of Body Composition and Physical Function in Older Adults With Obesity
Brief Title: Assessment of Body Composition and Physical Function
Acronym: Perform
Status: Completed | Type: Observational
Sponsor: Pennington Biomedical Research Center (Other)
Responsible Party: Principal Investigator, Candida Rebello, Assistant Professor, Pennington Biomedical Research Center
Other Study IDs: PBRC 2023-001
Record Dates: First submitted 2023-03-01; First posted 2023-03-27 (Actual); Results first posted 2024-07-30 (Actual); Last update posted 2024-07-30 (Actual); Status verified 2024-07

CONDITIONS: Body Composition; Physical Function
MeSH Terms: interventions — Hand Strength; Insulin

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Older Adults: Adults 60-80 years of age with body mass index > 30kg/m2
  Interventions: Other: Body Composition Assessment; Other: Modified Physical Performance Test; Other: Hand grip strength; Other: 6-minute walk test; Procedure: Measurement of blood glucose and insulin

INTERVENTIONS:
Other: Body Composition Assessment — Assessment of body composition using bioelectrical impedance analysis.
Other: Modified Physical Performance Test — A test of physical functioning
Other: Hand grip strength — A test of hand grip strength using a hand dynamometer.
Other: 6-minute walk test — Self-paced test of walking capacity.
Procedure: Measurement of blood glucose and insulin — Blood will be drawn for measurement of glucose and insulin.

SUMMARY:
Sarcopenia, which is the loss of muscle mass and strength or physical function, naturally occurs in aging. In sarcopenic obesity, growth of muscle mass and increments in strength do not parallel weight gain, and places older adults at increased risk of falls, fractures, physical disability, frailty, and mortality from too low muscle strength relative to body size. The goal of the study is to assess body composition and physical function in older adults with obesity.

DETAILED DESCRIPTION:
This is a cross-sectional study in 40 adults aged 60 to 80 years with obesity. Body composition, physical function, and insulin resistance will be measured. Subjects who satisfy the eligibility criteria and sign the informed consent will be enrolled. Subjects will complete an assessment of body composition by bioelectrical impedance analysis and tests of physical performance. Blood will be drawn for measurement of fasting glucose and insulin.

ELIGIBILITY:
Inclusion Criteria:

* Body mass index > 30kg/m2
* Age 60 - 80 years

Exclusion Criteria:

* self-reported history of diabetes, or cancer or significant cardiovascular or hepatic or renal disease or dysfunction.
* clinically significant gastrointestinal malabsorption syndromes such as chronic diarrhea, or celiac disease.

Ages: 60 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults aged 60 - 80 years with obesity.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2023-03-13 (Actual); Primary Completion 2023-06-01 (Actual); Study Completion 2023-06-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Candida J Rebello, Ph.D., Principal Investigator — Pennington Biomedical Research Center
Locations (1):
- Pennington Biomedical Research Center, Baton Rouge, Louisiana, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Gayoso-Diz P, Otero-Gonzalez A, Rodriguez-Alvarez MX, Gude F, Garcia F, De Francisco A, Quintela AG. Insulin resistance (HOMA-IR) cut-off values and the metabolic syndrome in a general adult population: effect of gender and age: EPIRCE cross-sectional study. BMC Endocr Disord. 2013 Oct 16;13:47. doi: 10.1186/1472-6823-13-47. PMID 24131857
- [Background] Ghasemi A, Tohidi M, Derakhshan A, Hasheminia M, Azizi F, Hadaegh F. Cut-off points of homeostasis model assessment of insulin resistance, beta-cell function, and fasting serum insulin to identify future type 2 diabetes: Tehran Lipid and Glucose Study. Acta Diabetol. 2015 Oct;52(5):905-15. doi: 10.1007/s00592-015-0730-3. Epub 2015 Mar 22. PMID 25794879

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Older Adults
Started | 40
Completed | 40
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Older Adults
Number analyzed (Participants) | 40
Age, Continuous [Mean (Standard Deviation); unit: years] | 67 (5.01)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 30
  Male | 10
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 9
  White | 30
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 40

OUTCOME MEASURES:

1. Primary Outcome: Fat Mass
Description: Measurement of fat mass
Time Frame: One day
Population: Older adults
Measure: Mean (Standard Deviation); unit: Kg
Arm/Group | Older Adults
Number analyzed (Participants) | 40
Kg | 44.71 (13.13)

2. Primary Outcome: Fat-free Mass
Description: Measurement of fat-free mass
Time Frame: One day
Population: Older adults
Measure: Mean (Standard Deviation); unit: Kg
Arm/Group | Older Adults
Number analyzed (Participants) | 40
Kg | 55.88 (12.08)

3. Primary Outcome: Modified Physical Performance Test
Description: Test for assessing physical performance. The scale ranges from 0 to 36 and higher score indicates a better outcome
Time Frame: One day
Population: Older adults
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Older Adults
Number analyzed (Participants) | 40
score on a scale | 30 (5.85)

4. Secondary Outcome: Hand Grip Strength
Description: Assessment of grip strength using a hand dynamometer
Time Frame: One day
Population: Average of the left- and right-hand grip strength measurement.
Measure: Mean (Standard Deviation); unit: kilograms
Arm/Group | Older Adults
Number analyzed (Participants) | 40
kilograms | 27.98 (9.36)

5. Secondary Outcome: 6-minute Walk Test
Description: Test of walking capacity assessed as distance covered in 6 minutes
Time Frame: One day
Measure: Mean (Standard Deviation); unit: Feet
Arm/Group | Older Adults
Number analyzed (Participants) | 40
Feet | 1375.25 (416.63)

6. Secondary Outcome: Homeostasis Model Assessment of Insulin Resistance (HOMA-IR)
Description: Assessment of insulin resistance from blood glucose and insulin. HOMA-IR was calculated as: fasting insulin (μU/mL) × fasting glucose (mmol/L)]/22.5 Higher scores indicate greater insulin resistance and a worse outcome. There is no theoretical minimum and/or maximum value for HOMA-IR. Studies have suggested a variety of values that vary based on factors such as gender and age. For example, a large epidemiologic study found that HOMA-IR score of 1.85 in women and 2.17 in men indicated insulin resistance. In another study, the HOMA-IR cut point was found to be 2.37 and 2.38 in 70-year old men and women respectively (see references).
Time Frame: One day
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Older Adults
Number analyzed (Participants) | 40
Score on a scale | 4.7 (3.4)

ADVERSE EVENTS:
Time Frame: Study was conducted over one visit.
Description: Adverse events were monitored and the presence or absence of an event was recorded during the conduct of the study visit.
Arm/Group | Older Adults
All-Cause Mortality (participants affected / at risk) | 0/40
Serious Adverse Events (participants affected / at risk) | 0/40
Other Adverse Events (participants affected / at risk) | 0/40

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-04-03): https://cdn.clinicaltrials.gov/large-docs/71/NCT05784571/Prot_SAP_000.pdf